CLINICAL TRIAL: NCT01016483
Title: Phase II Randomized Trial of MEK Inhibitor MSC1936369B or Placebo Combined With Gemcitabine in Metastatic Pancreas Cancer Subjects
Brief Title: Trial of Gemcitabine With or Without MSC1936369B in Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMR200066_003; 2009-011992-61 (EudraCT Number)
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: MEK inhibitor; cancer; pancreatic Adenocarcinoma; metastatic; chemo-naive; phase II
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — N-(2,3-dihydroxypropyl)-1-((2-fluoro-4-iodophenyl)amino)isonicotinamide; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Safety Run-in Part: Regimen 1 (Experimental): Subjects will receive pimasertib capsule orally once daily (qd) doses of 15, 30, 45, 68, 90, and 120 milligram (mg) on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
  Interventions: Drug: Pimasertib; Drug: Gemcitabine
- Safety Run-in Part: Regimen 2 (Experimental): Subjects will receive pimasertib capsule orally twice daily (bid) doses of 60 and 75 mg continuously for a 28-day cycle and gemcitabine 1000 mg/m^2 intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks) (bid - continuous regimen).
  Interventions: Drug: Pimasertib; Drug: Gemcitabine
- Phase II: Arm 1 (Gemcitabine + Placebo) (Active Comparator): Subjects will receive gemcitabine 1000 mg/m^2 IV infusion on for 30 minutes on Day 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1) then on Days 1, 8, and 15 of a 28-day cycle and placebo matched to pimasertib orally bid - continuous regimen.
  Interventions: Drug: Gemcitabine; Drug: Placebo
- Phase II: Arm 2 (Gemcitabine + Pimasertib) (Experimental): Subjects will receive gemcitabine 1000 mg/m^2 IV infusion for 30 minutes on Day 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1) then on Days 1, 8, and 15 of a 28-day cycle and pimasertib capsule orally bid - continuous regimen.
  Interventions: Drug: Pimasertib; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pimasertib
  Other Names: MSC1936369B (MEK Inhibitor)
  Arms: Phase II: Arm 2 (Gemcitabine + Pimasertib); Safety Run-in Part: Regimen 1; Safety Run-in Part: Regimen 2
Drug: Gemcitabine
Drug: Placebo
  Arms: Phase II: Arm 1 (Gemcitabine + Placebo)

SUMMARY:
The research trial is testing the experimental treatment MSC1936369B in combination with Gemcitabine, in subjects with metastatic pancreatic adenocarcinoma. The study will be run in two parts:

Safety Run-In: Will determine the Maximum Tolerated Dose (MTD) and the recommended Phase II dose of MSC1936369B, when combined with gemcitabine, in subjects with metastatic pancreatic adenocarcinoma.

Phase II: Will assess the anti-tumor activity of MSC1936369B combined with gemcitabine compared to gemcitabine alone as first line treatment in subjects with metastatic pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided signed informed consent. Fully understands requirements of the trial and willing to comply with all trial visits and assessments.
2. Histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas and availability of tumor sample.
3. Evidence of disease (not necessarily measurable disease). Complete tumor assessment including chest X ray, CT scan of abdomen and other scans as necessary to document all sites of disease performed within 28 days prior to trial entry/randomization.
4. Age ≥ 18 years.
5. Women of childbearing potential must have a negative blood pregnancy test at the screening visit. For the purposes of this trial, women of childbearing potential is defined as: "All female subjects after puberty unless they are post-menopausal for at least two years, are surgically sterile or are sexually inactive."
6. Female subjects of childbearing potential and male subjects with female partners of childbearing potential must be willing to avoid pregnancy by using an adequate method of contraception for 2 weeks prior to screening, during and four weeks after the last dose of trial medication. Adequate contraception is defined as two barrier methods, or one barrier method with a spermicide, or intrauterine device. The use of hormonal contraceptives should be avoided in female subjects of childbearing potential due to a possible drug-drug interaction.

Exclusion Criteria:

1. Bone marrow impairment as evidenced by hemoglobin less (<) 9.0 gram per deciliter (g/dL), neutrophil count < 1.5 x 10^9/ liter (L), platelets < 100 x 10^9/L.
2. Renal impairment as evidenced by serum creatinine > 1.5 x upper limit of normal (ULN), and/or calculated creatinine clearance < 60 mL/min.
3. Liver function abnormality as defined by total bilirubin > 1.5 x ULN, or aspartate aminotransferase/ alanine aminotransferase (AST/ALT) > 2.5 x ULN, for subjects with liver involvement AST/ALT > 5 x ULN.
4. Serum calcium > 1 x ULN.
5. History of central nervous system (CNS) metastases, unless subject has been previously treated for CNS metastases, is stable by CT scan without evidence of cerebral edema, and has no requirements for corticosteroids or anticonvulsants.
6. Eastern Cooperative Oncology Group Performance Status (ECOG PS) greater than 1.
7. Significant cardiac conduction abnormalities, including QT interval corrected for heart rate (QTc) prolongation of > 480 milliseconds (ms) and/or pacemaker.
8. Retinal degenerative disease (hereditary retinal degeneration or age-related macular degeneration), history of uveitis or history of retinal vein occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2009-11-30 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2015-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (2):
- For Recruiting Locations in the United States, please Contact U.S. Medical Information, Rockland, Massachusetts, United States
- For Recruiting Locations outside the United States, Please contact the Merck KGaA Communication Center, Darmstadt, Germany

REFERENCES:
- [Derived] Van Cutsem E, Hidalgo M, Canon JL, Macarulla T, Bazin I, Poddubskaya E, Manojlovic N, Radenkovic D, Verslype C, Raymond E, Cubillo A, Schueler A, Zhao C, Hammel P. Phase I/II trial of pimasertib plus gemcitabine in patients with metastatic pancreatic cancer. Int J Cancer. 2018 Oct 15;143(8):2053-2064. doi: 10.1002/ijc.31603. Epub 2018 Aug 9. PMID 29756206

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): Nov 2009/Jul 2013. Clinical data cut off: Dec 2013, Study completion date: April 2015
Groups:
- Safety Run-in Part: Regimen 1: Subjects received pimasertib capsule orally once daily (qd) doses of 15, 30, 45, 68, 90, and 120 milligram (mg) on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Safety Run-in Part: Regimen 2: Subjects received pimasertib capsule orally twice daily (bid) doses of 60 and 75 mg continuously for a 28-day cycle and gemcitabine 1000 mg/m^2 intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks) (bid continuous regimen).
- Phase II: Arm 1 (Gemcitabine + Placebo): Subjects received gemcitabine 1000 mg/m^2 IV infusion on for 30 minutes on Day 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1) then on Days 1, 8, and 15 of a 28-day cycle and placebo matched to pimasertib orally bid - continuous regimen. Subjects with disease progression in Arm 1 were allowed crossover to receive pimasertib capsule orally 60 mg bid - continuous regimen.
- Phase II: Arm 2 (Gemcitabine + Pimasertib): Subjects received gemcitabine 1000 mg/m^2 IV infusion on for 30 minutes on Day 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1) then on Days 1, 8, and 15 of a 28-day cycle and pimasertib capsule orally 60 mg bid - continuous regimen.
Period: Safety Run-in Part
Arm/Group | Safety Run-in Part: Regimen 1 | Safety Run-in Part: Regimen 2 | Phase II: Arm 1 (Gemcitabine + Placebo) | Phase II: Arm 2 (Gemcitabine + Pimasertib)
Started | 27 | 26 | 0 | 0
Completed | 27 | 26 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Safety Run-in Part: Regimen 1 | Safety Run-in Part: Regimen 2 | Phase II: Arm 1 (Gemcitabine + Placebo) | Phase II: Arm 2 (Gemcitabine + Pimasertib)
Started | 0 | 0 | 44 (Subjects presented as randomized (Intention-to-Treat [ITT] Analysis Set).) | 44 (Subjects presented as randomized (ITT Analysis Set).)
Treated (Safety Analysis Set [SAF]) | 0 | 0 | 42 (Subjects presented as treated (SAF).) | 45 (Subjects presented as treated (SAF).)
Completed | 0 | 0 | 44 | 44
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAF) analysis set for the safety run-in part included subjects who received at least 1 (non-zero) administration of trial medication (pimasertib or gemcitabine). For Phase II: Intention-to-treat (ITT) set included subjects who were randomized, as per Interactive Voice Response System (IVRS).
Groups:
- Safety Run-in Part: Regimen 2: Subjects received pimasertib capsule orally twice daily (bid) doses of 60 and 75 mg continuously for a 28-day cycle and gemcitabine 1000 mg/m^2 intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Total: Total of all reporting groups
Arm/Group | Safety Run-in Part: Regimen 1 | Safety Run-in Part: Regimen 2 | Phase II: Arm 1 (Gemcitabine + Placebo) | Phase II: Arm 2 (Gemcitabine + Pimasertib) | Total
Number analyzed (Participants) | 27 | 26 | 44 | 44 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 19 | 25 | 28 | 88
  >=65 years | 11 | 7 | 19 | 16 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 22 | 17 | 56
  Male | 18 | 18 | 22 | 27 | 85

OUTCOME MEASURES:

1. Primary Outcome: Safety Run-In Part: Number of Subjects With Dose Limiting Toxicities (DLTs)
Description: DLT using the National Cancer Institute Common Terminology Criteria for Adverse Events(CTCAE) v3.0,was defined as any of the following toxicities at any dose level and judged to be possibly or probably related to trial medication by the Investigator and/or the Sponsor and relevant for the combination treatment: Grade 3/more non-hematological toxicity excluding: Subjects with liver involvement: Grade 4 asymptomatic increases in liver function tests and subject without liver involvement: Grade 3 asymptomatic increases in liver function tests reversible within 7 days. Grade 3 vomiting encountered despite adequate therapy. Grade 3 diarrhea encountered despite adequate anti diarrhea therapy. Grade 4 neutropenia greater (>) 5 days duration or febrile neutropenia lasting for more than 1 day. Grade 4 thrombocytopenia > 1 day/Grade 3 with bleeding. Grade 4 anemia: Any treatment delay > 2 weeks due to drug-related adverse effects.
Time Frame: Up to 28 days in Cycle 1
Population: DLT analysis set included all subjects of safety run-in part who received any dose of pimasertib on at least 18 out of 20/25 out of 28 of the planned days on pimasertib & least 3 gemcitabine weekly infusions during first 28 days of treatment or experienced DLT during the 28 first days of treatment regardless of the amount of each drug received.
Measure: Number; unit: subjects
Groups:
- Safety Run-in Part Regimen 1: 15 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 15, mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Safety Run-in Part Regimen 1: 30 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 30, mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Safety Run-in Part Regimen 1: 45 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 45, mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Safety Run-in Part Regimen 1: 68 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 68, mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Safety Run-in Part Regimen 1: 90 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 90 mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Safety Run-in Part Regimen 1: 120 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 120 mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Safety Run-in Part Regimen 2: 60 mg: Subject received pimasertib capsule orally twice daily (bid) continuously for a 28-day cycle (60 mg bid - continuous regimen) and gemcitabine 1000 mg/m^2 intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1 = 8 weeks).
- Safety Run-in Part Regimen 2: 75 mg: Subject received pimasertib capsule orally twice daily (bid) continuously for a 28-day cycle (75 mg bid - continuous regimen) and gemcitabine 1000 mg/m^2 intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1 = 8 weeks).
Arm/Group | Safety Run-in Part Regimen 1: 15 mg | Safety Run-in Part Regimen 1: 30 mg | Safety Run-in Part Regimen 1: 45 mg | Safety Run-in Part Regimen 1: 68 mg | Safety Run-in Part Regimen 1: 90 mg | Safety Run-in Part Regimen 1: 120 mg | Safety Run-in Part Regimen 2: 60 mg | Safety Run-in Part Regimen 2: 75 mg
Number analyzed (Participants) | 3 | 2 | 3 | 2 | 2 | 8 | 10 | 9
subjects | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

2. Primary Outcome: Phase II: Progression-Free Survival (PFS) Time
Description: PFS was defined as the time from randomization to the first documentation of objective tumor progression (Complete Response (CR): Disappearance of all target lesions, Partial Response (PR): At least 30% decrease in the sum of the longest diameter of target lesions, taking as reference the sum of the longest diameter at baseline, Progressive Disease (PD): At least 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started, or the appearance of 1 or more new lesions and stable disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter since treatment started) or to death due to any cause, whichever occurred first. PFS calculated as (Months) = Date of first PD or death or censoring date minus date of randomization plus 1) divided by 30.4375.
Time Frame: From the time of randomization to every 8 weeks up to end of treatment (EOT) (6 years)
Population: Intent to Treat (ITT) analysis set included all subjects who had been randomized for the phase II part, as per the interactive voice response system (IVRS).
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase II: Arm 1: Subjects received gemcitabine 1000 mg/m^2 IV infusion on for 30 minutes on Day 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1) then on Days 1, 8, and 15 of a 28-day cycle and placebo orally bid - continuous regimen. Subjects with disease progression in Arm 1 were allowed crossover to receive pimasertib capsule orally 60 mg bid - continuous regimen.
- Phase II: Arm 2: Subjects received gemcitabine 1000 mg/m^2 IV infusion on for 30 minutes on Day 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1) then on Days 1, 8, and 15 of a 28-day cycle and pimasertib capsule orally 60 mg bid - continuous regimen.
Arm/Group | Phase II: Arm 1 | Phase II: Arm 2
Number analyzed (Participants) | 44 | 44
months | 2.83 [1.77 to 3.88] | 3.75 [2.63 to 5.09]

3. Secondary Outcome: Safety Run-In Part: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Permanent Treatment Discontinuation
Description: An adverse event (AE) was any untoward medical occurrence in a subjects who received study drug without regard to possibility of causal relationship. An serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. All AEs (serious and non-serious) except AEs recorded with an onset date prior to the first day of drug administration unless a worsening of the event was recorded after the first dosing date, in which case the event was counted as a TEAE. TEAEs include both SAEs and non-SAEs.
Time Frame: From the first dose of study drug administration until EOT (6 years)
Population: Safety analysis set (SAF) for the safety run-in part included all subjects who had received at least 1 administration of the trial medication (pimasertib or gemcitabine).
Measure: Number; unit: subjects
Arm/Group | Safety Run-in Part: Regimen 1 | Safety Run-in Part: Regimen 2
Number analyzed (Participants) | 27 | 26
subjects
  TEAEs | 27 | 26
  Serious TEAEs | 18 | 20
  Permanent treatment discontinuation of pimasertib | 12 | 16
  Permanent treatment discontinuation of gemcitabine | 14 | 15

4. Secondary Outcome: Safety Run-In Part: Maximum Concentration (Cmax) of Pimasertib (MSC1936369B), Gemcitabine (dFdC), and Gemcitabine Inactive Metabolite 2',2'-Difluorodeoxyuridine (dFdU) for Regimen 1
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: Pharmacokinetic set (PKS) of the safety run in part included subjects who had received at least the first dose of both drugs (i.e., gemcitabine and pimasertib), and provided PK samples as per the protocol for at least 24 hours following first dosing on Day1. Here "n" signifies number of subjects evaluable for each category at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Regimen 1: 15 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 15, mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Regimen 1: 30 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 30, mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Regimen 1: 45 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 45, mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Regimen 1: 68 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 68, mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Regimen 1: 90 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 90 mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Regimen 1: 120 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 120 mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
Arm/Group | Regimen 1: 15 mg | Regimen 1: 30 mg | Regimen 1: 45 mg | Regimen 1: 68 mg | Regimen 1: 90 mg | Regimen 1: 120 mg
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 11
nanogram per milliliter (ng/mL)
  MSC1936369B on Days 1 (n=4,3,3,3,3,11) | 32.3 (107.5) | 131.0 (32.9) | 205.8 (30.0) | 151.3 (40.1) | 485.3 (58.7) | 484.3 (39.8)
  MSC1936369B on Days 22 (n= 3,3,3,2,3,10) | 29.6 (39.8) | 174.2 (29.6) | 261.8 (52.0) | 212.5 (16.9) | 409.1 (44.1) | 252.9 (477.0)
  Gemcitabine (dFdC) on Day 1 (n=4,3,3,3,3,11) | 69540.5 (1729.4) | 21207.3 (21.0) | 17759.9 (34.1) | 29762.1 (76.7) | 15606.3 (23.1) | 23880.7 (83.8)
  Gemcitabine (dFdC) on Day 22 (n= 2,3,3,2,3,9) | 24115.8 (71.9) | 11799.7 (167.7) | 181.9 (39158542.7) | 163196.2 (3183.3) | 669.5 (3278825923) | 23207.2 (99.5)
  Metabolite (dFdU) on Day 1 (n= 4,3,3,3,3,11) | 29359.8 (8.5) | 33171.6 (21.2) | 34868.9 (12.8) | 33804.4 (16.7) | 37786.4 (13.6) | 34038.7 (29.7)
  Metabolite (dFdU) on Day 22 (n= 2,3,3,2,3,10) | 29677.6 (3.0) | 38265.2 (54.3) | 10569.2 (449.2) | 32869.2 (8.7) | 17135.0 (227.5) | 21077.5 (179.5)

5. Secondary Outcome: Safety Run-In Part: Time to Reach Maximum Concentration (Tmax) of Pimasertib (MSC1936369B), Gemcitabine (dFdC), and Gemcitabine Inactive Metabolite 2',2'-Difluorodeoxyuridine (dFdU): Regimen 1
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: PKS set of the safety run in part included subjects who had received at least the first dose of both drugs (i.e., gemcitabine and pimasertib), and provided PK samples as per the protocol for at least 24 hours following first dosing on Day 1. Here "n" signifies number of subjects evaluable for each category at specified time point.
Measure: Median (Full Range); unit: hours
Groups:
- Regimen 1: 15 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 15 mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Regimen 1: 68 mg: Subjects received pimasertib orally once daily (qd) 5-days-on / 2-days-off, continuously (Days 1 to 5, 8 to 12, 15 to 19, 22 to 26, and so on) dose of 68 mg and gemcitabine 1000 milligram per square meter (mg/m^2) 30 minutes intravenous (IV) infusion on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1 = 8 weeks) then on Days 1, 8, and 15 of a 28-day cycle.
- Regimen 1: 90 mg: Subjects received pimasertib orally once daily (qd) 5-days-on / 2-days-off, continuously (Days 1 to 5, 8 to 12, 15 to 19, 22 to 26, and so on) dose of 90 mg and gemcitabine 1000 milligram per square meter (mg/m^2) 30 minutes intravenous (IV) infusion on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1 = 8 weeks) then on Days 1, 8, and 15 of a 28-day cycle.
- Regimen 1: 120 mg: Subjects received pimasertib orally once daily (qd) 5-days-on / 2-days-off, continuously (Days 1 to 5, 8 to 12, 15 to 19, 22 to 26, and so on) dose of 120 mg and gemcitabine 1000 milligram per square meter (mg/m^2) 30 minutes intravenous (IV) infusion on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1 = 8 weeks) then on Days 1, 8, and 15 of a 28-day cycle.
Arm/Group | Regimen 1: 15 mg | Regimen 1: 30 mg | Regimen 1: 45 mg | Regimen 1: 68 mg | Regimen 1: 90 mg | Regimen 1: 120 mg
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 11
hours
  Tmax: MSC1936369B on Day 1 (n= 4,3,3,3,3,11) | 1.250 [1.00 to 1.50] | 1.000 [1.00 to 2.50] | 1.533 [1.00 to 2.00] | 2.000 [0.67 to 8.00] | 1.083 [1.00 to 2.00] | 1.500 [0.50 to 4.00]
  Tmax: MSC1936369B on Day 22 (n= 3,3,3 2,3,10) | 2.017 [1.28 to 4.00] | 1.000 [0.50 to 2.50] | 1.000 [0.50 to 1.58] | 1.750 [1.00 to 2.50] | 1.500 [1.00 to 1.75] | 2.000 [0.83 to 8.00]
  Tmax: Gemcitabine (dFdC) on Day 1 (n=4,3,3,3,3,11) | 0.38 [0.25 to 0.50] | 0.50 [0.25 to 0.50] | 0.25 [0.25 to 0.50] | 0.25 [0.25 to 1.17] | 0.25 [0.25 to 0.38] | 0.27 [0.25 to 0.75]
  Tmax: Gemcitabine (dFdC) on Day 22 (n=2,3,3,2,3,9) | 0.42 [0.33 to 0.50] | 0.50 [0.50 to 1.58] | 0.53 [0.25 to 2.00] | 1.04 [1.00 to 1.08] | 0.25 [0.23 to 24.00] | 0.50 [0.25 to 0.75]
  Tmax: Metabolite (dFdU) on Day 1 (n=4,3,3,3,3,11) | 0.64 [0.50 to 1.00] | 0.50 [0.50 to 0.75] | 0.50 [0.50 to 0.77] | 0.75 [0.67 to 1.00] | 0.50 [0.38 to 0.50] | 0.50 [0.25 to 0.75]
  Tmax: Metabolite (dFdU) on Day 22 (n=2,3,3,2,3,10 | 0.54 [0.33 to 0.75] | 0.75 [0.50 to 1.58] | 1.00 [0.73 to 2.00] | 0.67 [0.33 to 1.00] | 0.75 [0.50 to 24.00] | 0.75 [0.00 to 1.00]

6. Secondary Outcome: Safety Run-In Part: Time to Reach Apparent Terminal Half-Life (t1/2) of Pimasertib (MSC1936369B), Gemcitabine (dFdC), and Gemcitabine Inactive Metabolite 2',2'-Difluorodeoxyuridine (dFdU): Regimen 1
Description: Plasma decay half-life was the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Groups:
- Regimen 1: 30 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 30 mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Regimen 1: 45 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 45 mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Regimen 1: 68 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 68 mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
Arm/Group | Regimen 1: 15 mg | Regimen 1: 30 mg | Regimen 1: 45 mg | Regimen 1: 68 mg | Regimen 1: 90 mg | Regimen 1: 120 mg
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 11
hours
  t1/2: MSC1936369B on Day 1 (n=4,3,3,2,3,11) | 4.008 [2.539 to 6.131] | 3.807 [3.373 to 6.648] | 3.833 [3.612 to 6.477] | 4.232 [3.382 to 5.083] | 5.036 [4.361 to 5.120] | 4.580 [3.394 to 6.938]
  t1/2: MSC1936369B on Day 22 (n=2,2,3,2,3,8) | 8.660 [4.709 to 12.61] | 6.100 [4.878 to 7.322] | 3.254 [3.048 to 6.999] | 5.744 [3.829 to 7.658] | 3.162 [2.903 to 6.341] | 4.825 [2.829 to 8.642]
  t1/2: Gemcitabine (dFdC) on Day 1 (n=4,3,3,3,3,11) | 4.274 [2.100 to 7.519] | 2.461 [1.239 to 6.821] | 2.421 [0.7070 to 5.709] | 5.327 [5.148 to 5.338] | 8.940 [5.565 to 9.982] | 6.242 [0.8913 to 11.90]
  t1/2: Gemcitabine (dFdC) on Day 22 (n=2,2,1,2,2,9) | 7.449 [6.032 to 8.866] | 4.553 [2.403 to 6.702] | 0.9152 [0.9152 to 0.9152] | 4.493 [2.721 to 6.266] | 8.213 [6.665 to 9.762] | 4.680 [0.8685 to 8.490]
  t1/2: Metabolite (dFdU) on Day 1 (n=4,3,3,3,3,11) | 8.956 [8.129 to 14.68] | 10.49 [4.336 to 10.70] | 9.836 [9.383 to 14.69] | 11.52 [9.344 to 12.36] | 8.349 [7.191 to 9.551] | 10.93 [8.802 to 15.48]
  t1/2: Metabolite (dFdU) on Day 22(n=2,2,2,2,2,10) | 7.731 [6.978 to 8.483] | 8.925 [8.299 to 9.552] | 8.843 [5.427 to 12.26] | 11.14 [9.119 to 13.17] | 10.21 [6.782 to 13.64] | 12.17 [3.468 to 211.2]

7. Secondary Outcome: Safety Run-In Part: Area Under Curve (AUC: 0 to Infinity) of Pimasertib (MSC1936369B), Gemcitabine (dFdC), and Gemcitabine Inactive Metabolite 2',2'-Difluorodeoxyuridine (dFdU): Regimen 1
Description: AUC:0 to infinity was a measure of the serum concentration of the drug over time. It was used to characterize drug absorption.
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1 of Cycle 1 for MSC1936369B, 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1 for Gemcitabine
Population: PKS of the safety run in part included subjects who had received at least the first dose of both drugs (i.e., gemcitabine and pimasertib), and provided PK samples as per the protocol for at least 24 hours following first dosing on Day 1. Here "n" signifies number of subjects evaluable for each category at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Regimen 1:15 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 15 mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
- Regimen1: 120 mg: Subjects received pimasertib capsule orally once daily (qd) doses of 120 mg on Day 1, 2, 3, 4, 5, 8, 9, 10, 11, 12, 15,16, 17, 18, 19, 22, 23, 24, 25, 26 and gemcitabine 1000 milligram per square meter (mg/m^2) intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (1 Cycle = 8 weeks).
Arm/Group | Regimen 1:15 mg | Regimen 1: 30 mg | Regimen 1: 45 mg | Regimen 1: 68 mg | Regimen 1: 90 mg | Regimen1: 120 mg
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 11
hour*nanogram per milliliter (h*ng/mL)
  AUC: MSC1936369B on Day 1 (n=4,3,3,3,3,11) | 162.8 (25.3) | 516.3 (32.9) | 881.1 (37.1) | 774.8 (58.9) | 1729.9 (32.3) | 2175.1 (53.0)
  AUC: Gemcitabine (dFdC) on Day 1(n=4,3,3,3,3,11) | 29536.1 (473.4) | 13536.5 (40.4) | 10053.3 (24.6) | 18956.0 (37.2) | 8178.4 (28.7) | 11680.1 (59.0)
  AUC: Gemcitabine (dFdC) on Day 22(n=2,2,1,2,2,9) | 10828.0 (93.8) | 12019.6 (29.5) | 9093.2 (NA) — Data for Geometric Coefficient of Variation was not estimable as only one subject was analyzed. | 76448.7 (466.6) | 9604.8 (11.9) | 10598.0 (66.7)
  AUC: Metabolite (dFdU) on Day 1 (n=4,3,3,3,3,11) | 245795.5 (10.8) | 228032.9 (27.6) | 276968.3 (28.9) | 259816.2 (9.2) | 239902.9 (27.1) | 240293.8 (15.0)
  AUC: Metabolite (dFdU) on Day 22 (n=2,2,2,2,2,10) | 190952.6 (9.3) | 376280.5 (13.0) | 217930.8 (70.4) | 327424.8 (2.0) | 248496.4 (5.2) | 247430.7 (29.2)

8. Secondary Outcome: Safety Run-In Part: Apparent Oral Clearance (CL/f) of Pimasertib (MSC1936369B): Regimen 1
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) was influenced by the fraction of the dose absorbed.
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Regimen 1:15 mg | Regimen 1: 30 mg | Regimen 1: 45 mg | Regimen 1: 68 mg | Regimen 1: 90 mg | Regimen 1: 120 mg
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 11
Liter per hour (L/h)
  CL/f: MSC1936369B on Day 1 (n=4,3,3,2,3,11) | 92.152 (25.3) | 58.104 (32.9) | 51.072 (37.1) | 87.765 (58.9) | 52.025 (32.3) | 55.171 (53.0)
  CL/f: MSC1936369B on Day 22 (n=2,2,3,2,3,9) | 74.143 (43.6) | 42.484 (31.2) | 44.579 (23.1) | 56.502 (7.5) | 50.873 (59.6) | 55.723 (57.8)

9. Secondary Outcome: Safety Run-In Part: Total Clearance (CL) of Gemcitabine: Regimen 1
Description: Clearance of a drug was a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: PKS set of the safety run in part included subjects who had received at least the first dose of both drugs (i.e., gemcitabine and pimasertib), and provided PK samples as per the protocol for at least 24 hours following first dosing on Day 1. Here "n" signifies those subjects who were evaluable at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Regimen 1: 15 mg | Regimen 1: 30 mg | Regimen 1: 45 mg | Regimen 1: 68 mg | Regimen 1: 90 mg | Regimen 1: 120 mg
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 11
liter/hour
  CL: Gemcitabine on Day 1 (n=4,3,3,3,3,11) | 60.537 (483.4) | 133.88 (45.1) | 190.52 (26.0) | 95.96 (47.7) | 210.25 (27.9) | 151.93 (54.7)
  CL: Gemcitabine on Day 22 (n=2,2,1,2,2,9) | 163.37 (93.7) | 156.93 (20.1) | 190.69 (NA) — Data for Geometric Coefficient of Variation was not estimable as only one subject was analyzed. | 25.123 (431.2) | 183.97 (11.6) | 164.6 (71.7)

10. Secondary Outcome: Safety Run-In Part: Oral Volume of Distribution (V/f) of Pimasertib (MSC1936369B): Regimen 1
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Regimen 1: 15 mg | Regimen 1: 30 mg | Regimen 1: 45 mg | Regimen 1: 68 mg | Regimen 1: 90 mg | Regimen 1: 120 mg
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 11
liter
  V/f: MSC1936369B on Day 1 (n=4,3,3,2,3,11) | 528.62 (63.1) | 369.12 (5.0) | 329.80 (28.4) | 524.96 (26.2) | 362.29 (34.0) | 367.25 (50.5)
  V/f: MSC1936369B on Day 22 (n=2,2,3,2,3,8) | 824.33 (156.8) | 366.30 (1.8) | 264.31 (43.8) | 441.40 (43.4) | 284.42 (35.1) | 414.38 (66.8)

11. Secondary Outcome: Safety Run-In Part: Apparent Volume of Distribution (V) of Gemcitabine: Regimen 1
Description: Apparent volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Regimen 1: 15 mg | Regimen 1: 30 mg | Regimen 1: 45 mg | Regimen 1: 68 mg | Regimen 1: 90 mg | Regimen 1: 120 mg
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 11
liter
  V: Gemcitabine (dFdC) on Day 1 (n= 4,3,3,3,3,11) | 359.55 (635.6) | 531.23 (64.7) | 587.64 (206.3) | 729.65 (46.3) | 2402.1 (59.5) | 1270.1 (82.0)
  V: Gemcitabine (dFdC) on Day 22 (n=2,2,1,2,2,9) | 1723.6 (55.9) | 908.50 (56.5) | 251.79 (NA) — Data for Geometric Coefficient of Variation was not estimable as only one subject was analyzed. | 149.65 (1453.7) | 2140.8 (15.5) | 805.15 (138.0)

12. Secondary Outcome: Safety Run-In Part: Levels of Pharmacodynamic (Pd) Markers (Phosphorylated- Extracellular Signal-Regulated Kinase (ERK) in Peripheral Blood Mononuclear Cells [PBMCs]): Regimen 1
Description: ERK phosphoprotein in peripheral blood monocytes (PBMCs) was analyzed from blood samples of all subjects in the SAF analysis set (safety-run part) only.
Time Frame: pre-dose on Day 1, 2, 22 of Cycle 1; post-dose on Day 1, 22 of Cycle 1
Population: Pharmacodynamic population included SAF analysis set for the safety run-in part include all subjects who received at least 1 (non-zero) administration of the trial medication (pimasertib or gemcitabine). Here "n" signifies those subjects who were evaluable at the specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: Fluorescence Intensity
Arm/Group | Regimen 1:15 mg | Regimen 1: 30 mg | Regimen 1: 45 mg | Regimen 1: 68 mg | Regimen 1: 90 mg | Regimen1: 120 mg
Number analyzed (Participants) | 3 | 2 | 2 | 3 | 3 | 7
Fluorescence Intensity
  Cycle 1 Day 1 Pre-dose (n=3,2,2,3,3,7) | 5.389 (0.797) | 6.476 (0.997) | 4.767 (0.114) | 6.509 (2.240) | 4.608 (0.197) | 4.229 (1.719)
  Cycle 1 Day 1 Post-dose (n=3,2,2,3,2,6) | 1.611 (0.537) | 2.061 (0.825) | 0.837 (0.149) | 3.881 (5.387) | 1.059 (0.042) | 0.946 (0.248)
  Cycle 1 Day 2 Pre-dose (n=3,2,1,2,2,6) | 4.818 (0.808) | 6.719 (2.835) | 3.902 (NA) — Data for standard deviation was not estimable as only one subject was analyzed. | 2.768 (0.330) | 4.874 (2.119) | 3.636 (1.755)
  Cycle 1 Day 22 Pre-dose (n=2,1,2,1,3,5) | 5.242 (0.210) | 6.000 (NA) — Data for standard deviation was not estimable as only one subject was analyzed. | 1.978 (2.539) | 8.653 (NA) — Data for standard deviation was not estimable as only one subject was analyzed. | 4.252 (1.259) | 3.453 (0.860)
  Cycle 1 Day 22 Post-dose (n=0,0,0,0,2) | NA (NA) — No subjects were evaluable at the specified time point hence the parameter was not analyzed. | NA (NA) — No subjects were evaluable at the specified time point hence the parameter was not analyzed. | NA (NA) — No subjects were evaluable at the specified time point hence the parameter was not analyzed. | NA (NA) — No subjects were evaluable at the specified time point hence the parameter was not analyzed. | NA (NA) — No subjects were evaluable at the specified time point hence the parameter was not analyzed. | 4.130 (1.772)

13. Secondary Outcome: Safety Run-In Part: Maximum Concentration (Cmax) of Pimasertib (MSC1936369B), Gemcitabine (dFdC), Gemcitabine Inactive Metabolite 2',2'-Difluorodeoxyuridine (dFdU): Regimen 2
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Regimen 2: 60 mg: Subject received pimasertib capsule orally twice daily (bid) continuously for a 28-day cycle (60 mg bid - continuous regimen) and gemcitabine 1000 mg/m^2 intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1 = 8 weeks).
- Regimen 2: 75 mg: Subject received pimasertib capsule orally twice daily (bid) continuously for a 28-day cycle (75 mg bid - continuous regimen) and gemcitabine 1000 mg/m^2 intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1 = 8 weeks).
Arm/Group | Regimen 2: 60 mg | Regimen 2: 75 mg
Number analyzed (Participants) | 12 | 14
nanogram per milliliter (ng/mL)
  MSC1936369B on Day 1 (n= 12,13) | 175.7 (65.0) | 345.5 (52.8)
  MSC1936369B on Day 22 (n=10,9) | 228.2 (59.0) | 244.8 (31.9)
  Gemcitabine (dFdC) on Day 1 (n=11,14) | 27849.2 (344.0) | 17663.9 (173.3)
  Gemcitabine (dFdC) on Day 22 (n=9,4) | 21589.7 (118.8) | 18733.4 (88.6)
  Gemcitabine Metabolite (dFdU) on Day 1 (n=11, 10) | 33033.3 (11.8) | 31623.9 (25.4)
  Gemcitabine Metabolite (dFdU) on Day 22 (n=10,5) | 13455.5 (546.0) | 18298.7 (247.7)

14. Secondary Outcome: Safety Run-In Part: Area Under Curve (AUC:0 to Infinity) of Pimasertib (MSC1936369B), Gemcitabine (dFdC), and Gemcitabine Inactive Metabolite 2',2'-Difluorodeoxyuridine (dFdU) Regimen 2
Description: AUC:0 to infinity is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Groups:
- Regimen 1: 75 mg: Subject received pimasertib capsule orally twice daily (bid) continuously for a 28-day cycle (75 mg bid - continuous regimen) and gemcitabine 1000 mg/m^2 intravenous (IV) infusion for 30 minutes on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1 = 8 weeks).
Arm/Group | Regimen 2: 60 mg | Regimen 1: 75 mg
Number analyzed (Participants) | 12 | 14
hour*nanogram per milliliter (h*ng/mL)
  AUC: MSC1936369B on Day 1 (n= 10, 11) | 704.3 (69.4) | 1427.0 (30.0)
  AUC: Gemcitabine (dFdC) on Day 1 (n= 11, 14) | 11932.0 (343.0) | 8065.5 (176.2)
  AUC: Gemcitabine (dFdC) on Day 22 (n= 9, 4) | 10719.1 (84.9) | 10102.3 (72.0)
  AUC: Metabolite (dFdU) on Day 1 (n= 11, 13) | 189007.0 (40.6) | 234934.8 (29.9)
  AUC: Metabolite (dFdU) on Day 22 (n= 10, 5) | 177504.5 (171.5) | 256714.9 (37.3)

15. Secondary Outcome: Safety Run-In Part: Time to Reach Maximum Concentration (Tmax) of Pimasertib (MSC1936369B), Gemcitabine (dFdC), and Gemcitabine Inactive Metabolite 2',2'-Difluorodeoxyuridine (dFdU): Regimen 2
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: PKS set of the safety run in part included subjects who had received at least the first dose of both drugs (i.e., gemcitabine and pimasertib), and provided PK samples as per the protocol for at least 24 hours following first dosing on Day 1.Here "n" signifies number of subjects evaluable for each category at specified time point.
Measure: Median (Full Range); unit: hours
Arm/Group | Regimen 2: 60 mg | Regimen 2: 75 mg
Number analyzed (Participants) | 12 | 14
hours
  Tmax: MSC1936369B on Day 1 (n=12,13) | 2.000 [0.50 to 3.98] | 1.583 [0.50 to 7.98]
  Tmax: MSC1936369B on Day 22 (n=10,9) | 1.500 [0.25 to 4.40] | 2.000 [0.58 to 4.00]
  Tmax: Gemcitabine (dFdC) on Day 1 (n=11,14) | 0.50 [0.25 to 0.73] | 0.38 [0.25 to 0.75]
  Tmax: Gemcitabine (dFdC) on Day 22 (n=9,4) | 0.25 [0.00 to 0.50] | 0.25 [0.25 to 0.50]
  Tmax: Metabolite (dFdU) on Day 1 (n=11,13) | 0.67 [0.50 to 0.75] | 0.67 [0.25 to 1.00]
  Tmax: Metabolite (dFdU) on Day 22 (n=10,5) | 0.50 [0.00 to 2.00] | 0.50 [0.50 to 0.75]

16. Secondary Outcome: Safety Run-In Part: Time to Reach Apparent Terminal Half-Life (t1/2) of Pimasertib (MSC1936369B), Gemcitabine (dFdC), and Gemcitabine Inactive Metabolite 2',2'-Difluorodeoxyuridine (dFdU): Regimen 2
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Regimen 2: 60 mg | Regimen 2: 75 mg
Number analyzed (Participants) | 12 | 14
hours
  t1/2: MSC1936369B on Day 1 (n=10,11) | 2.757 [2.183 to 3.557] | 2.603 [1.775 to 4.910]
  t1/2: MSC1936369B on Day 22 (n=8,5) | 3.425 [2.584 to 10.60] | 3.188 [2.296 to 4.617]
  t1/2: Gemcitabine (dFdC) on Day 1 (n=11,14) | 5.258 [0.796 to 8.757] | 5.376 [0.6681 to 11.64]
  t1/2: Gemcitabine (dFdC) on Day 22 (n=9,4) | 5.522 [3.759 to 11.45] | 5.249 [0.3198 to 9.505]
  t1/2: Metabolite (dFdU) on Day 1 (n=11,13) | 9.471 [6.559 to 13.10] | 10.26 [7.123 to 12.92]
  t1/2: Metabolite (dFdU) on Day 22 (n=10,5) | 10.68 [6.543 to 441.9] | 13.58 [7.575 to 17.535]

17. Secondary Outcome: Safety Run-In Part: Apparent Oral Clearance (CL/f) of Pimasertib (MSC1936369B): Regimen 2
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed.
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/H)
Arm/Group | Regimen 2: 60 mg | Regimen 2: 75 mg
Number analyzed (Participants) | 12 | 14
Liter per hour (L/H)
  CL/f: MSC1936369B on Day 1 (n=10,11) | 85.186 (69.4) | 52.558 (30.0)
  CL/f: MSC1936369B on Day 22 (n=8,5) | 70.163 (63.2) | 68.312 (24.9)

18. Secondary Outcome: Safety Run-In Part: Total Clearance (CL) of Gemcitabine: Regimen 2
Description: as for outcome 9
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Groups:
- Regimen 2: 60 mg: Subjects received pimasertib orally twice daily (bid) continuously without a break for a 28-day cycle (60 mg bid - continuous regimen) and gemcitabine 1000 milligram per square meter (mg/m^2) 30 minutes intravenous (IV) infusion on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1 = 8 weeks) then on Days 1, 8, and 15 of a 28-day cycle.
- Regimen 2: 75 mg: Subjects received pimasertib orally twice daily (bid) continuously without a break for a 28-day cycle (75 mg bid - continuous regimen) and gemcitabine 1000 milligram per square meter (mg/m^2) 30 minutes intravenous (IV) infusion on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1 = 8 weeks) then on Days 1, 8, and 15 of a 28-day cycle.
Arm/Group | Regimen 2: 60 mg | Regimen 2: 75 mg
Number analyzed (Participants) | 12 | 14
liter/hour
  CL: Gemcitabine on Day 1 (n=11, 14) | 145.65 (363.2) | 221.46 (186.0)
  CL: Gemcitabine on Day 22 (n=9, 4) | 164.68 (81.4) | 183.85 (73.5)

19. Secondary Outcome: Safety Run-In Part: Apparent Volume of Distribution (V) of Gemcitabine: Regimen 2
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug.
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Regimen 2: 60 mg | Regimen 2: 75 mg
Number analyzed (Participants) | 12 | 14
liter
  V: Gemcitabine on Day 1 (n=11,14) | 716.12 (343.3) | 1059.0 (196.6)
  V: Gemcitabine on Day 22 (n=9,4) | 1590.8 (120.5) | 801.90 (130.3)

20. Secondary Outcome: Safety Run-In Part: Oral Volume of Distribution (V/f) of Pimasertib (MSC1936369B): Regimen 2
Description: as for outcome 10
Time Frame: 0 hour (pre-dose), 0.5, 1, 1.5, 2, 2.5, 4, 8, 12, 24 (post-dose) on Day 1, 22 of Cycle 1
Population: PKS set of the safety run in part included subjects who had received at least the first dose of both drugs (i.e. gemcitabine and pimasertib), and provided PK samples as per the protocol for at least 24 hours following first dosing on Day 1. Here "n" signifies number of subjects evaluable for each category at specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Regimen 2: 60 mg | Regimen 2: 75 mg
Number analyzed (Participants) | 12 | 14
liter
  V/f: MSC1936369B on Day 1 (n= 10,11) | 335.56 (66.3) | 213.24 (37.7)
  V/f: MSC1936369B on Day 22 (n=8,5) | 389.56 (47.1) | 319.02 (35.5)

21. Secondary Outcome: Safety Run-In Part: Levels of Pharmacodynamic (Pd) Markers (Phosphorylated- Extracellular Signal-Regulated Kinase (ERK) in Peripheral Blood Mononuclear Cells [PBMCs]): Regimen 2
Description: as for outcome 12
Time Frame: pre-dose on Day 1, 2, 22 of Cycle 1; post-dose on Day 1, 22 of Cycle 1
Population: Pharmacodynamic population included SAF analysis set for the safety run-in part include all subjects who received at least 1 (non-zero) administration of the trial medication (pimasertib or gemcitabine). Here "n" signifies those subjects who were evaluable at the specified time point for each arm respectively.
Measure: Mean (Standard Deviation); unit: Fluorescence Intensity
Arm/Group | Regimen 2: 60 mg | Regimen 2: 75 mg
Number analyzed (Participants) | 7 | 4
Fluorescence Intensity
  Cycle 1 Day 1 Pre-dose (n=7,4) | 6.081 (0.827) | 5.874 (2.239)
  Cycle 1 Day 1 Post-dose (n=5,3) | 1.520 (0.109) | 1.048 (0.155)
  Cycle 1 Day 2 Pre-dose (n=7,3) | 3.877 (2.099) | 2.263 (0.593)
  Cycle 1 Day 22 Pre-dose (n=6,2) | 2.728 (0.818) | 2.295 (0.510)
  Cycle 1 Day 22 Post-dose (n=3,1) | 1.443 (0.458) | 1.111 (NA) — Data for standard deviation was not estimable as only one subject was analyzed.

22. Secondary Outcome: Phase II: Number of Subjects With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs Leading to Permanent Treatment Discontinuation
Description: An AE was any untoward medical occurrence in a subject who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. All AEs (serious and non-serious) except AEs recorded with an onset date prior to the first day of drug administration unless a worsening of the event was recorded after the first dosing date, in which case the event was counted as a TEAE. TEAEs include both SAEs and non-SAEs.
Time Frame: From the first dose of study drug administration until EOT (6 years)
Population: SAF for the Phase II included all subjects who had received at least 1 administration of the trial medication Gemcitabine or Placebo if the subject is in the gemcitabine + Placebo treatment arm (Arm 1) and MSC1936369B or gemcitabine in the MSC1936369B + gemcitabine treatment arm (Arm 2).
Measure: Number; unit: subjects
Arm/Group | Phase II: Arm 1 | Phase II: Arm 2
Number analyzed (Participants) | 42 | 45
subjects
  TEAEs | 40 | 45
  Serious TEAEs | 28 | 35
  TEAEs Leading to Treatment Discontinuation | 10 | 21

23. Secondary Outcome: Phase II: Percentage of Subjects With Best Overall Response (BOR)
Description: Best overall response was defined as the presence of at least one complete response (CR), partial response (PR) or Stable Disease (SD) (using RECIST v1.0) during treatment. CR: Disappearance of all target lesions, PR: At least 30% decrease in the sum of the longest diameter of target lesions, taking as reference the sum of the longest diameter at baseline and SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter since treatment started.
Time Frame: Baseline, every 8 weeks up to end of treatment (EOT i.e. 6 years)
Population: ITT analysis set included all subjects who had been randomized for the phase II part, as per the interactive voice response system (IVRS).
Measure: Number; unit: percentage of subjects
Arm/Group | Phase II: Arm 1 | Phase II: Arm 2
Number analyzed (Participants) | 44 | 44
percentage of subjects
  CR | 0 | 0
  PR | 9.1 | 9.1
  SD | 36.4 | 50.0
  PD | 29.5 | 20.5
  Missing | 25 | 20.5

24. Secondary Outcome: Phase II: Percentage of Subjects With Clinical Benefit
Description: Clinical Benefit was defined as the presence of at least one CR, PR or Stable Disease (SD) (using RECIST v1.0) during treatment. CR: Disappearance of all target lesions, PR: At least 30% decrease in the sum of the longest diameter of target lesions, taking as reference the sum of the longest diameter at baseline and SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of the longest diameter since treatment started.
Time Frame: Baseline, every 8 weeks up to end of treatment (EOT i.e. 6 years)
Population: as for outcome 23
Measure: Number; unit: percentage of subjects
Arm/Group | Phase II: Arm 1 | Phase II: Arm 2
Number analyzed (Participants) | 44 | 44
percentage of subjects | 45.5 | 59.1

25. Secondary Outcome: Phase II: Time to Progression (TTP)
Description: Time to progression (TTP) is defined as the time (in months) from the randomization date to the date of progression prior to the start of any subsequent therapy for the primary disease, as reported and documented by the Investigator (i.e. radiological progression per RECIST).
Time Frame: From randomization every 8 weeks up to EOT (6 years)
Population: as for outcome 23
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Arm 1 | Phase II: Arm 2
Number analyzed (Participants) | 44 | 44
months | 3.78 [1.87 to 5.55] | 5.09 [3.75 to 6.47]

26. Secondary Outcome: Phase II: Overall Survival (OS) Time
Description: Overall survival (OS) time is defined as the time (in months) from randomization to death.
Time Frame: Baseline, every 8 weeks up to EOT (6 years)
Population: as for outcome 23
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Arm 1 | Phase II: Arm 2
Number analyzed (Participants) | 44 | 44
months | 6.64 [5.06 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to limited number of events. | 9.33 [3.71 to NA] — Upper limit of 95% Confidence Interval (CI) was not estimable due to limited number of events.

27. Secondary Outcome: Phase II: Absorption Rate Constant (ka) of Pimasertib (MSC1936369B)
Time Frame: Baseline, every 8 weeks up to EOT (6 years)
Population: As per change in planned analysis, there was reduction of PK investigations for the phase II part of the trial, removal of PK sampling for gemcitabine and its metabolites and replacement of intense sampling with a sparse sampling scheme for pimasertib, thus the outcome measure was not analyzed.
Arm/Group | Phase II: Arm 1 | Phase II: Arm 2
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Phase II: Clearance From Central Compartment (CL/f) and Intercompartmental Clearance (Q/f) of Pimasertib (MSC1936369B)
Time Frame: Baseline, every 8 weeks up to EOT (6 years)
Population: as for outcome 27
Arm/Group | Phase II: Arm 1 | Phase II: Arm 2
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Phase II: Volume of Central Compartment (V1/f) and Volume of Peripheral Compartment (V2/f) of Pimasertib (MSC1936369B)
Time Frame: Baseline, every 8 weeks up to EOT (6 years)
Population: as for outcome 27
Arm/Group | Phase II: Arm 1 | Phase II: Arm 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration until EOT (6 years)
Description: Adverse Events were collected for SAF. SAF for safety run-in part included all subjects who had received at least 1 administration of trial medication (pimasertib or gemcitabine). SAF for Phase II included all subjects who had received at least 1 administration of trial medication Gemcitabine or Placebo if subject is in gemcitabine + Placebo arm (Arm 1) or at least 1 administration of trial medication MSC1936369B or gemcitabine if subject is in MSC1936369B + gemcitabine arm (Arm 2).
Groups:
- Phase II: Arm 1: Subjects received gemcitabine 1000 mg/m^2 for 30 minutes IV infusion on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1) then on Days 1, 8, and 15 of a 28-day cycle and placebo orally bid - continuous regimen. Subjects with disease progression in Arm 1 were allowed crossover to receive pimasertib orally 60 mg bid - continuous regimen.
- Phase II: Arm 2: Subjects received gemcitabine 1000 mg/m^2 for 30 minutes IV infusion on Days 1, 8, 15, 22, 29, 36, and 43 followed by a 1-week rest (Cycle 1) then on Days 1, 8, and 15 of a 28-day cycle and pimasertib orally 60 mg bid - continuous regimen.
Arm/Group | Safety Run-in Part: Regimen 1 | Safety Run-in Part: Regimen 2 | Phase II: Arm 1 | Phase II: Arm 2
Serious Adverse Events (participants affected / at risk) | 18/27 | 20/26 | 28/42 | 35/45
Other Adverse Events (participants affected / at risk) | 27/27 | 26/26 | 39/42 | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Part: Regimen 1 (N=27) | Safety Run-in Part: Regimen 2 (N=26) | Phase II: Arm 1 (N=42) | Phase II: Arm 2 (N=45)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukaemoid reaction (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 3
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 4
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Chorioretinopathy (Eye disorders) | 0 | 1 | 0 | 0
Macular detachment (Eye disorders) | 0 | 0 | 0 | 1
Retinal Vein Occlusion (Eye disorders) | 0 | 2 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 2 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 4
Asthenia (General disorders) | 2 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 1 | 2
Disease progression (General disorders) | 1 | 0 | 5 | 4
Fatigue (General disorders) | 0 | 0 | 0 | 2
General physical health deterioration (General disorders) | 2 | 2 | 1 | 3
Malaise (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Oedema Peripheral (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 6 | 5 | 5
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 3 | 1 | 2 | 2
Cholangitis Acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 3 | 1
Jaundice extrahepatic obstructive (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cystitis klebsiella (Infections and infestations) | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Enterobacter sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 0 | 1 | 0
Hepatitis c (Infections and infestations) | 0 | 1 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 2
Pulmonary sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 3 | 5
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 4 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Coma (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Palliative Care (Surgical and medical procedures) | 1 | 0 | 0 | 0
Capillary Leak Syndrome (Vascular disorders) | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Part: Regimen 1 (N=27) | Safety Run-in Part: Regimen 2 (N=26) | Phase II: Arm 1 (N=42) | Phase II: Arm 2 (N=45)
Neutropenia (Blood and lymphatic system disorders) | 14 | 6 | 17 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 13 | 9 | 16
Anaemia (Blood and lymphatic system disorders) | 10 | 9 | 8 | 13
Leukopenia (Blood and lymphatic system disorders) | 5 | 4 | 6 | 4
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 3
Retinal detachment (Eye disorders) | 10 | 14 | 1 | 10
Macular degeneration (Eye disorders) | 4 | 3 | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 3 | 1 | 4
Visual impairment (Eye disorders) | 5 | 2 | 0 | 4
Eyelid oedema (Eye disorders) | 1 | 4 | 0 | 3
Vision blurred (Eye disorders) | 2 | 2 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 14 | 19 | 8 | 20
Abdominal pain (Gastrointestinal disorders) | 9 | 4 | 11 | 7
Constipation (Gastrointestinal disorders) | 9 | 6 | 8 | 8
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2 | 7 | 4
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 1 | 3
Nausea (Gastrointestinal disorders) | 16 | 15 | 15 | 23
Vomiting (Gastrointestinal disorders) | 13 | 12 | 11 | 22
Stomatitis (Gastrointestinal disorders) | 12 | 12 | 4 | 15
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 2 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 3
Fatigue (General disorders) | 15 | 5 | 17 | 17
Oedema peripheral (General disorders) | 14 | 15 | 8 | 22
Pyrexia (General disorders) | 14 | 11 | 12 | 17
Asthenia (General disorders) | 8 | 13 | 6 | 9
Gamma-glutamyltransferase increased (Investigations) | 0 | 3 | 7 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 9
Alanine aminotransferase increased (Investigations) | 6 | 4 | 4 | 4
Aspartate aminotransferase increased (Investigations) | 4 | 5 | 3 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 6 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 3 | 3 | 4
Platelet count decreased (Investigations) | 0 | 0 | 1 | 5
Weight decreased (Investigations) | 3 | 2 | 4 | 1
Ejection fraction decreased (Investigations) | 2 | 2 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 10 | 11 | 9 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 2 | 2 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 6 | 3 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 5 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 5 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 3 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 6 | 4 | 20
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 4 | 1 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 7 | 2 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 3
Hypotension (Vascular disorders) | 0 | 0 | 1 | 4
Normochromic Normocytic Anaemia (Blood and lymphatic system disorders) | 5 | 0 | 0 | 1
Anaemia of Chronic Disease (Blood and lymphatic system disorders) | 2 | 2 | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 2 | 2 | 4
Aphthous Stomatitis (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 9 | 9 | 0 | 1
Exfoliative Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 1
Pain of Skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 3 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4 | 2 | 1
Haemoglobin Decreased (Investigations) | 3 | 2 | 0 | 2
Transaminases Increased (Investigations) | 1 | 2 | 1 | 1
Dysgeusia (Nervous system disorders) | 6 | 4 | 2 | 2
Headache (Nervous system disorders) | 6 | 1 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 3 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 7
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 1 | 2
Insomnia (Psychiatric disorders) | 3 | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 2 | 1 | 2
Disorientation (Psychiatric disorders) | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 5 | 2 | 2 | 1
Capillary leak syndrome (Vascular disorders) | 0 | 3 | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Haemoglobinaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Dilatation ventricular (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 2 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 2 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Scotoma (Eye disorders) | 4 | 5 | 0 | 0
Papilloedema (Eye disorders) | 2 | 0 | 0 | 0
Colour blindness acquired (Eye disorders) | 1 | 1 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0
Retinal pigment epitheliopathy (Eye disorders) | 1 | 0 | 0 | 0
Retinal vascular disorder (Eye disorders) | 1 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 1 | 4 | 0 | 1
Chorioretinopathy (Eye disorders) | 0 | 2 | 0 | 1
Macular oedema (Eye disorders) | 0 | 2 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0
Cystoid macular oedema (Eye disorders) | 0 | 1 | 0 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 2 | 0
Ocular discomfort (Eye disorders) | 0 | 1 | 0 | 0
Ocular toxicity (Eye disorders) | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 1 | 0 | 0
Retinal exudates (Eye disorders) | 0 | 1 | 0 | 0
Retinoschisis (Eye disorders) | 0 | 1 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0
Macular detachment (Eye disorders) | 0 | 0 | 0 | 7
Detachment of macular retinal pigment epithelium (Eye disorders) | 0 | 0 | 0 | 2
Arteriosclerotic retinopathy (Eye disorders) | 0 | 0 | 1 | 0
Cataract nuclear (Eye disorders) | 0 | 0 | 0 | 1
Eye disorder (Eye disorders) | 0 | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 1
Eye oedema (Eye disorders) | 0 | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1
Photopsia (Eye disorders) | 0 | 0 | 0 | 1
Retinal disorder (Eye disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Oral submucosal fibrosis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Palatal oedema (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enlarged uvula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Aerophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 5 | 2 | 1 | 0
Oedema (General disorders) | 2 | 1 | 0 | 1
Chills (General disorders) | 1 | 2 | 3 | 1
Face oedema (General disorders) | 1 | 2 | 1 | 2
Feeling cold (General disorders) | 1 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 3 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 1 | 2
Hypothermia (General disorders) | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Device failure (General disorders) | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0
Injection site haematoma (General disorders) | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 3 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 4
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
BRONCHITIS (Infections and infestations) | 3 | 1 | 0 | 1
Lung infection (Infections and infestations) | 2 | 0 | 0 | 0
Paronychia (Infections and infestations) | 2 | 1 | 0 | 1
Escherichia infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 0
Oral fungal infection (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 2
Pneumonia klebsiella (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 3 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 1 | 1
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 0
Pneumocystis jiroveci infection (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis klebsiella (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Open wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Postoperative hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0
Visual field tests abnormal (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0 | 0
Blood sodium increased (Investigations) | 0 | 1 | 0 | 0
Transferrin saturation decreased (Investigations) | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 3 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 2
Blood albumin increased (Investigations) | 0 | 0 | 0 | 2
Blood iron decreased (Investigations) | 0 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1
Blood creatine increased (Investigations) | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 0
Red blood cell count decreased (Investigations) | 0 | 0 | 0 | 1
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Aphonia (Nervous system disorders) | 1 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 1
Restless leg syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 0
Allodynia (Nervous system disorders) | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 2
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 2
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 1 | 0 | 2
Visual field defect (Nervous system disorders) | 0 | 1 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 2
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal infarct (Renal and urinary disorders) | 0 | 0 | 1 | 0
Epididymal tenderness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Prostatism (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Sunburn (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 1
Phlebitis (Vascular disorders) | 1 | 1 | 1 | 0
Lymphoedema (Vascular disorders) | 0 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other